CLINICAL TRIAL: NCT07016243
Title: Correlation Between Deficits in ROM Recovery of the Knee Operated With PTG and Difficulty in Dorsiflexing the Tibio-tarsal Joint.NODORSIFLEX-IN-PTG
Brief Title: Correlation Between Deficits in Knee ROM Recovery and Difficulty in Dorsiflexing the Tibio-tarsal Joint in Patients Undergoing Total Knee Replacement Surgery.
Acronym: NODORSIFLEX
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 0003043-01/03/2025
Record Dates: First submitted 2025-05-16; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Articulation Disorders
MeSH Terms: conditions — Articulation Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To demonstrate that the deficit in dorsiflexion-tibia-talar joint range of motion can have an effect on the knee operated by arthroplasty by limiting full extension and, in general, the recovery of a full range of motion.

DETAILED DESCRIPTION:
The study is of a prospective, prognostic, observational nature and involves all patients who are candidates for admission to the Rizzoli Orthopaedic Institute for primary knee replacement surgery, recruited in the Orthopaedics department and subsequently followed in the Rehabilitation Medicine department of the DRS. The recruited patients will be subjected to pre-operative measurement of the ankle ROM; if they present a limitation of the same, they will be included in the exposed group, alternatively they will be included in the non-exposed group.

ELIGIBILITY:
Inclusion Criteria:•

* Patients who are candidates for primary total knee replacement surgery aged 65 to 85 years;
* Patients who have provided informed consent Exclusion Criteria:•
* Patients with known neurological pathologies
* Severe joint deformations such as previous ankle surgery (arthrodesis, ankle prosthesis) congenital malformations (cavus equinus, clubfoot)
* Severe fractures that have compromised the joint
* Traumatic events affecting the lower limb that occurred less than 12 months
* Non-ambulatory patients in the preoperative period

Ages: 65 Years to 85 Years | Sex: All
Age Groups: Older Adult
Study Population: To demonstrate in a Physical Medicine and Rehabilitation department that the deficit in dorsiflexion-tibia-talar joint range of motion can have an effect on the knee operated on with arthroplasty by limiting complete extension and, in general, the recovery of a complete range of motion.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of knee joint range of motion (ROM). | In our study, the joint excursion measurements of the t-t and knee will be taken by the physiotherapists involved in the study with the patient lying in a supine position on a bed, they will be taken pre-operatively (T0) i.e. before the knee arthroplasty
  The study is of a prospective, prognostic, observational nature and involves all patients who are candidates for admission to the Rizzoli Orthopedic Institute for primary knee replacement surgery, recruited in the Orthopedics department and subsequently followed in the Rehabilitation Medicine department of the DRS. The recruited patients will be subjected to pre-operative measurement of the ankle ROM; if they present a limitation of the same, they will be included in the exposed group, alternatively they will be included in the non-exposed group.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Tornatore, Principal Investigator — Istituto Ortopedico Rizzoli - Dipartimento Sicilia
Locations (1):
- Istituto Ortopedico Rizzoli Dipartimento Sicilia, Bagheria, Palermo, Italy